CLINICAL TRIAL: NCT01722851
Title: Novel Breast Cancer Biomarkers and Their Use for Guiding and Monitoring Response to Chemotherapy
Brief Title: Circulating miRNAs.
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 10-11
Record Dates: First submitted 2012-10-24; First posted 2012-11-07 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Newly Diagnosed Breast Cancer; Recurrent Breast Cancer
Keywords: Breast Cancer; miRNAs; Newly diagnosed; Recurrent
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Cohort 1: All newly diagnosed breast cancer patients who are scheduled to undergo neoadjuvant chemotherapy
- Cohort 2: All breast cancer patients who present with metastatic disease, disease recurrence or progression, who are commencing up-front chemotherapy ± hormonal therapy
- Cohort 3: All breast cancer patient who present with metastatic disease who are commencing hormonal therapy only.

SUMMARY:
To identify a panel of circulating miRNA markers which could help identify those breast cancer patients who are most likely to respond well to neoadjuvant and adjuvant chemotherapy, and indeed serve as an overall prognostic factor and stratify patients into risk categories which would further guide their management. Similarly, the investigators aim to identify a panel of circulating miRNA markers which could monitor patient's response to chemotherapy and hormonal therapies. Ideally a suitable panel of markers would show significant changes in expression level in good-responders whilst little or no change would be observed in miRNA expression in non-responders.

DETAILED DESCRIPTION:
Primary Objectives:

1. To identify a panel of miRNAs, detectable in the circulation, which are altered in breast cancer patients
2. To identify specific combinations of miRNAs ('signatures') which associate with breast cancer intrinsic subtypes, and thereby could aid in prognostication and treatment planning on an individual patient basis.

Secondary Objective:

1. To determine if systemic miRNA analysis can be used as a biomarker for monitoring response to chemotherapy, in the neoadjuvant setting and in patients who present with breast cancer recurrence and are treated with upfront chemotherapy and/or hormonal therapy.

   This is a prospective cohort studies, involving three study cohorts:

   Cohort 1: All newly diagnosed breast cancer patients who are scheduled to undergo neoadjuvant chemotherapy.

   Cohort 2: All breast cancer patients who present with metastatic disease, disease recurrence or progression, who are commencing up-front chemotherapy +/- hormonal therapy.

   Cohort 3: All breast cancer patients who present with metastatic disease who are commencing hormonal therapy only.

   Blood Sample

   Blood Sampling - Cohort 1:

   - Blood sample 1: at presentation before commencing neoadjuvant treatment.

   - Blood sample 2: midway through their chemotherapy treatment (after 2nd cycle if they are enrolled in a 4 cycle regimen, or after 4th cycle if they are prescribed an 8 week regimen).

   - Blood sample 3: post-chemotherapy (before surgery as applicable).

   - Blood sample 4: 2 to 4 weeks after surgery, or 2 to 4 weeks post 3rd blood sampling if patients do not undergo surgery.

   - Blood sample 5: once during follow-up of 12 to 18 months after surgery or 12 to 18 months post 3rd blood sampling if patients do not undergo surgery.

   Blood Sampling - Cohort 2:

   - Pre-treatment blood sample: at presentation before commencing treatment.

   - On study blood samples: taken at monthly (± 1 week) intervals for a period of 6 months from date of pre-treatment blood sample, despite whether the patient is on treatment or completed treatment.

   On study blood sample 1: 1 month (± 1 week) from date of pre-treatment blood sample

   On study blood sample 2: 2 months (± 1 week) from date of pre- treatment blood sample

   On study blood sample 3: 3 months (± 1 week) from date of pre-treatment blood sample

   On study blood sample 4: 4 months (± 1 week) from date of pre-treatment blood sample

   On study blood sample 5: 5 months (± 1 week) from date of pre-treatment blood sample

   On study blood sample 6: 6 months (± 1 week) from date of pre-treatment blood sample

   - End of study blood sample: once during follow-up of 12 to 18 months from date of pre-treatment blood sample or at the time of disease progression.

   Blood Sampling - Cohort 3:

   - Pre-treatment blood sample: at presentation before commencing treatment.

   - On study blood samples: taken at the following time points despite whether the patient is on treatment or completed treatment.

   On study blood sample 1: 3 months (± 2 weeks) from date of pre-treatment blood sample On study blood sample 2: 6 months (± 2 weeks) from date of pre-treatment blood sample On study blood sample 3: 12 months (± 2 weeks) from date of pre-treatment blood sample

   - End of study blood sample: 18 months (± 2 weeks) from date of pre-treatment blood sample or at the time of disease progression.

   Blood samples will be processed for miRNA analysis, which involves:

1. Lysis using Trizol 2. RNA isolation 3. Assessing concentration and integrity of RNA using Nanodrop spectrophotometry 4. cDNA synthesis (using miRNA specific stem loop primers) 5. PCR amplification and relative quantification (using miRNA specific probes)

ELIGIBILITY:
Inclusion Criteria

1. Patient must meet the criteria for either:

   Cohort 1: All patients with a new diagnosis of breast cancer, who are destined to undergo neoadjuvant chemotherapy.

   OR Cohort 2: All breast cancer patients who present with metastatic disease, disease recurrence or progression who will receive up-front chemotherapy ± hormonal therapy.

   OR Cohort 3: All breast cancer patient who present with metastatic disease who are commencing hormonal therapy only.
2. Patients must be aged 18 years or over.
3. Patients must be able to give written informed consent.

Exclusion Criteria

All patients, who do not fulfil the inclusion criteria mentioned above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators aim to study two populations of breast cancer patients:
  1. Patients undergoing neoadjuvant chemotherapy for breast cancer at tertiary referral breast cancer centres in Ireland.
     For GUH only: Additionally,investigators wish to evaluate miRNA expression levels in patients' diagnostic core biopsies.
  2. Investigators also wish to study the same panel of miRNAs in patients who present with disease recurrence or disease progression, and who are commenced on systemic therapies (hormonal and/or chemotherapy).
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Relationship between changes in a patients circulating miRNA expression levels over the course of their systemic therapy, and their response to that treatment. | Up to week 66-92
  For cohort 1, a patient's response to treatment will be determined using 3 standard parameters: clinical, radiological and pathological responses.
  For cohort 2 and 3, a patient's response to treatment will be evaluated using RECIST criteria version 1.1." For cohort 1, a patient's response to treatment will be determined using 3 standard parameters: clinical, radiological and pathological responses.
  For cohort 2 and 3, a patient's response to treatment will be evaluated using RECIST criteria version 1.1."
Correlation of systemic miRNA levels with standard biomarkers of response | Up to week 66-92
  Standard bio markers of response include serum CEA and Ca15-3 levels

SECONDARY OUTCOMES:
Relationship between circulating miRNA profiles and patients' intrinsic subtype of breast cancer | Up to week 66-92
Relationship between miRNA expression levels and other existing clinicopathological parameters. | Up to week 66-92
  Other existing clinicopathological parameters include: ER, PR and HER2 status, stage of disease,histological grade and size of the tumour, and the Nottingham Prognostic Index.

CONTACTS AND LOCATIONS:
Locations (7):
- Ireland (7):
  - Bon Secours Hospital, Cork
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Galway, Galway
  - Letterkenny General Hospital, Letterkenny
  - Sligo General Hospital, Sligo
  - Midlands Regional Hospital Tullamore, Tullamore

REFERENCES:
- [Derived] Davey MG, McGuire A, Casey MC, Waldron RM, Paganga M, Holian E, Newell J, Heneghan HM, McDermott AM, Keane MM, Lowery AJ, Miller N, Kerin MJ. Evaluating the Role of Circulating MicroRNAs in Predicting Long-Term Survival Outcomes in Breast Cancer: A Prospective, Multicenter Clinical Trial. J Am Coll Surg. 2023 Feb 1;236(2):317-327. doi: 10.1097/XCS.0000000000000465. Epub 2022 Nov 2. PMID 36648259
- [Derived] Davey MG, Casey MC, McGuire A, Waldron RM, Paganga M, Holian E, Newell J, Heneghan HM, McDermott AM, Keane MM, Lowery AJ, Miller N, Kerin MJ. Evaluating the Role of Circulating MicroRNAs to Aid Therapeutic Decision Making for Neoadjuvant Chemotherapy in Breast Cancer: A Prospective, Multicenter Clinical Trial. Ann Surg. 2022 Nov 1;276(5):905-912. doi: 10.1097/SLA.0000000000005613. Epub 2022 Jul 25. PMID 35876391